CLINICAL TRIAL: NCT03969368
Title: Randomized Trial of rPMS Pelvic Floor Stimulation Device Compared With Pelvic Floor Exercises for Treatment of Urinary Incontinence
Brief Title: rPMS Compared With Pelvic Floor Exercises for Treatment of Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BTL Industries Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BTL-099-U2
Record Dates: First submitted 2019-05-28; First posted 2019-05-31 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Treatment Group (Experimental): Treatment with the investigational device - rPMS
  Interventions: Device: rPMS device
- Control Group (Active Comparator): Control group
  Interventions: Procedure: Pelvic floor muscle training

INTERVENTIONS:
Device: rPMS device — Pelvic floor muscle contractions will be induced by the rPMS device.
  Arms: Treatment Group
Procedure: Pelvic floor muscle training — Control group will undergo a pelvic floor muscle training
  Arms: Control Group

SUMMARY:
This study will compare the clinical efficacy and safety between rPMS device and pelvic floor exercises for the treatment of urinary incontinence. The subjects will be enrolled and assigned into two study groups - active and control group. Subjects will be required to complete six (6) treatment visits and five follow-up visits - 1, 3, 6, 9 and 12 months after the final treatment.

ELIGIBILITY:
Inclusion Criteria:

* Female aged 25-70 years
* Suffers from specific types of UI - Stress Urinary Incontinence (SUI), Urge Urinary Incontinence (UUI) and/or Mixed Urinary Incontinence (MUI)
* Voluntarily signed informed consent form
* Subjects willing and able to abstain from partaking in any treatment of urinary incontinence other than the study procedure
* Subjects currently undergoing any treatment for stress, urge and/or mixed urinary incontinence, have to undergo a two-week wash-out period before start of the study

Exclusion Criteria:

* Use of Botox® in the bladder or pelvic muscles in the last year
* Use of Interstim® or similar device for the treatment of UI
* Suffers from other types of urinary incontinence other than SUI, UUI, MUI
* Pelvic organ prolapse grade 2 and higher
* Pronounced lesions of the pudendus nerve during clinical neurophysiological examination
* Currently lactating
* Cardiac pacemakers
* Implanted defibrillators and/or neurostimulators
* Electronic implants
* Metal implants, including copper IUD
* Drug pumps
* Hemorrhagic conditions
* Anticoagulation therapy
* Fever
* Pregnancy
* Following recent surgical procedures when muscle contraction may disrupt the healing process
* Application over areas of the skin which lack normal sensation
* Any disorders that the Investigator deems would interfere with study endpoints or subject safety

Ages: 25 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-07-23 (Actual); Study Completion 2022-06-23 (Actual)

PRIMARY OUTCOMES:
Evaluation of quality of life improvement using the UDI-6 questionnaire | 13 months
  Evaluation of change in UDI-6 score before and after the study treatment in both study groups. Decrease of the score will be considered as an improvement.
Evaluation of incontinence episodes using Bladder diary | 13 months
  Evaluation of change in incontinence episodes before and after the study treatment in both study groups.
Evaluation of quality of life improvement using the ICIQ-LUTSqol questionnaire | 13 months
  Evaluation of change in ICIQ-LUTSqol score before and after the study treatment in both study groups. Decrease of the score will be considered as an improvement.
Evaluation of quality of life improvement using the Pad Usage Questionnaire | 13 months
  Evaluation of change in Pad Usage Questionnaire before and after the study treatment in both study groups. Decrease in number of used pads will be considered as an improvement.
Evaluation of pelvic floor muscle strength | 13 months
  Evaluation of pelvic floor muscle strength with measurement of voluntary contraction in both study groups.

SECONDARY OUTCOMES:
Subject Satisfaction evaluation | 13 months
  Qualitative analysis of subject's opinion using a questionnaire. Subjects will be asked to describe the change and their satisfaction after the study treatment.
Therapy comfort evaluation | 1 month
  Evaluation of therapy comfort after each treatment or training session using the questionnaire.
Safety evaluation | 13 months
  Incidence of adverse events (AE) associated with study device will be followed.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Boston Urogyn, Wellesley, Massachusetts
  - Center for Urogynecology and Reconstructive Surgery, Somerset, New Jersey
  - The Female Pelvic Health Center, Newtown, Pennsylvania
  - The Female Pelvic Medicine Institute, Richmond, Virginia